CLINICAL TRIAL: NCT04436094
Title: Soft Tissue Outcomes Of Badly Broken-Down Teeth Treated With Orthodontic Extrusion Compared With Immediate Implant Placement: A Randomized Controlled Trial
Brief Title: Soft Tissue Outcomes Of Badly Broken-Down Teeth Treated With Orthodontic Extrusion Compared With Immediate Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moustafa Osama Shehata, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22042020
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Broken Teeth
MeSH Terms: conditions — Tooth Fractures | interventions — Orthodontic Extrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthodontic extrusion (Experimental): An orthodontic attachment will be bonded to the core of the experimental tooth. Orthodontic brackets "American Orthodontics Roth prescription. 0.022" slot" will be bonded to the adjacent teeth. A passive rectangular stainless steel wire (0.016X0.022") will be inserted in the adjacent teeth with a step down and a coil at the site of the experimental tooth.
  Orthodontic extrusion will start using a light overlay wire of 0.012" NiTi and then continued by elastic chains/ threads extending between the attachment on the tooth and the stabilizing wire. The patient is followed up for appliance activation every 3-4 weeks and extrusion is performed until an adequate ferrule effect of 2 mm is present all around the tooth circumference (in addition to the biologic width). So the extrusion is completed when the tooth is 4-4.5 mm from the alveolar bone crest as judged by periapical radiographs.
  Interventions: Procedure: Orthodontic extrusion
- Immediate implant placement (Active Comparator): The patient is anaesthetized. Atraumatic extraction of the badly broken down teeth will be performed using peroiotome. Luxation should be done mesiodistally and not buccolingually, to avoid damaging the buccal plate. After tooth removal, a curette is used to confirm that the location of the buccal plate is intact. Standard drilling procedures are performed according to the manufacturer's instructions. Then the implant is placed in the prepared site. Temporization should be done using composite 3M Filtek Z250 XT material. Finally, a porcelain fused to zirconia crown will be performed.
  Interventions: Procedure: Immediate implant placement

INTERVENTIONS:
Procedure: Orthodontic extrusion — An orthodontic attachment will be bonded to the core of the experimental tooth. Orthodontic brackets "American Orthodontics Roth prescription. 0.022" slot" will be bonded to the adjacent teeth. A passive rectangular stainless steel wire (0.016X0.022") will be inserted in the adjacent teeth with a step down and a coil at the site of the experimental tooth.
  Orthodontic extrusion will start using a light overlay wire of 0.012" NiTi and then continued by elastic chains/ threads extending between the attachment on the tooth and the stabilizing wire. The patient is followed up for appliance activation every 3-4 weeks and extrusion is performed until an adequate ferrule effect of 2 mm is present all around the tooth circumference (in addition to the biologic width). So the extrusion is completed when the tooth is 4-4.5 mm from the alveolar bone crest as judged by periapical radiographs.
  Arms: Orthodontic extrusion
Procedure: Immediate implant placement — The patient is anaesthetized. Atraumatic extraction of the badly broken down teeth will be performed using peroiotome. Luxation should be done mesiodistally and not buccolingually, to avoid damaging the buccal plate. After tooth removal, a curette is used to confirm that the location of the buccal plate is intact. Standard drilling procedures are performed according to the manufacturer's instructions. Then the implant is placed in the prepared site. Temporization should be done using composite 3M Filtek Z250 XT material. Finally, a porcelain fused to zirconia crown will be performed.
  Arms: Immediate implant placement

SUMMARY:
Many patients suffer from tooth substance loss as a result of fracture or decay of teeth situated in the esthetic zone. This might commonly occur with car accidents, sport injuries, falls or even fistfights.

For those patients, most of the crown is lost and only the root remains, so there is no enough ferrule in order to restore the tooth with a crown.

The most common treatment for those patients is immediate single-tooth implant. However, some problems may arise such as: high treatment expenses, the need for bone augmentation, the refill of the papilla to its normal position may be questionable in some implant cases, young growing patients, apprehensive patients, dental facilities and rural areas lacking cone beam computed tomography (CBCT) machines.

Accordingly, orthodontic extrusion may be an alternative attempt to preserve the tooth by traction of the remaining root to create a sufficient ferrule effect to restore the tooth.

ELIGIBILITY:
Inclusion Criteria:

* Patients at 20-40 years old and have no history of periodontal disease. (periodontally healthy patients).
* Single rooted teeth with adjacent intact or restored neighboring teeth, more than one tooth may be included in the same arch.
* More than 1:1 crown root ratio, so that the C/R is 1:1 after extrusion and restoration.
* Presence of intact adjacent teeth.

Exclusion Criteria:

* Badly broken-down teeth with active signs of infection.
* Teeth with vertical root fracture.
* Teeth with severely tapered roots..
* Diabetic patients, assessed by measuring glycosylated hemoglobin (HbA1c). Patients with an HbA1c level greater than 8 will be excluded.
* Potentially uncooperative patients who are not willing to go through the proposed interventions (patients who will refuse to undergo orthodontic treatment).
* Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day).
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems, emotional instability, and unrealistic esthetic demands.
* History of radiation therapy to the head and neck, or bone augmentation to implant site.
* Labial cortical bone fenestration diagnosed from CBCT.
* Bruxism.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Soft tissue outcome | 12 months
  Pink esthetic score: 0-1-2 scoring system, 0 being the lowest, 2 being the highest value

SECONDARY OUTCOMES:
Survival | 12 months
  Tooth and Implant survival

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa O Shehata, B.D.S., Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bastone EB, Freer TJ, McNamara JR. Epidemiology of dental trauma: a review of the literature. Aust Dent J. 2000 Mar;45(1):2-9. doi: 10.1111/j.1834-7819.2000.tb00234.x. PMID 10846265
- [Background] Juloski J, Radovic I, Goracci C, Vulicevic ZR, Ferrari M. Ferrule effect: a literature review. J Endod. 2012 Jan;38(1):11-9. doi: 10.1016/j.joen.2011.09.024. Epub 2011 Nov 13. PMID 22152612
- [Background] Olsburgh S, Jacoby T, Krejci I. Crown fractures in the permanent dentition: pulpal and restorative considerations. Dent Traumatol. 2002 Jun;18(3):103-15. doi: 10.1034/j.1600-9657.2002.00004.x. PMID 12110103
- [Background] Rosenberg ES, Cho SC, Garber DA. Crown lengthening revisited. Compend Contin Educ Dent. 1999 Jun;20(6):527-32, 534, 536-8 passim; quiz 542. PMID 10650366
- [Background] Grossmann Y, Sadan A. The prosthodontic concept of crown-to-root ratio: a review of the literature. J Prosthet Dent. 2005 Jun;93(6):559-62. doi: 10.1016/j.prosdent.2005.03.006. PMID 15942617
- [Background] Alsahhaf A, Att W. Orthodontic extrusion for pre-implant site enhancement: Principles and clinical guidelines. J Prosthodont Res. 2016 Jul;60(3):145-55. doi: 10.1016/j.jpor.2016.02.004. Epub 2016 Mar 12. PMID 26979626
- [Background] Elkhadem A, Mickan S, Richards D. Adverse events of surgical extrusion in treatment for crown-root and cervical root fractures: a systematic review of case series/reports. Dent Traumatol. 2014 Feb;30(1):1-14. doi: 10.1111/edt.12051. Epub 2013 Jun 25. PMID 23796195
- [Background] Yuan LT, Duan DM, Tan L, Wang XJ, Wu LA. Treatment for a complicated crown-root fracture with intentional replantation: a case report with a 3.5-year follow up. Dent Traumatol. 2013 Dec;29(6):474-8. doi: 10.1111/j.1600-9657.2012.01130.x. Epub 2012 Mar 27. PMID 22453056
- [Background] Malmgren O, Malmgren B, Frykholm A. Rapid orthodontic extrusion of crown root and cervical root fractured teeth. Endod Dent Traumatol. 1991 Apr;7(2):49-54. doi: 10.1111/j.1600-9657.1991.tb00183.x. PMID 1782893
- [Background] Schwartz-Arad D, Chaushu G. Placement of implants into fresh extraction sites: 4 to 7 years retrospective evaluation of 95 immediate implants. J Periodontol. 1997 Nov;68(11):1110-6. doi: 10.1902/jop.1997.68.11.1110. PMID 9407405
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Smith DE, Zarb GA. Criteria for success of osseointegrated endosseous implants. J Prosthet Dent. 1989 Nov;62(5):567-72. doi: 10.1016/0022-3913(89)90081-4. PMID 2691661
- [Background] Albrektsson T, Zarb GA. Determinants of correct clinical reporting. Int J Prosthodont. 1998 Sep-Oct;11(5):517-21. No abstract available. PMID 9922743
- [Background] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Background] Annibali S, Bignozzi I, La Monaca G, Cristalli MP. Usefulness of the aesthetic result as a success criterion for implant therapy: a review. Clin Implant Dent Relat Res. 2012 Mar;14(1):3-40. doi: 10.1111/j.1708-8208.2009.00234.x. Epub 2009 Aug 6. PMID 19673953
- [Background] Meijer HJ, Stellingsma K, Meijndert L, Raghoebar GM. A new index for rating aesthetics of implant-supported single crowns and adjacent soft tissues--the Implant Crown Aesthetic Index. Clin Oral Implants Res. 2005 Dec;16(6):645-9. doi: 10.1111/j.1600-0501.2005.01128.x. PMID 16307570
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- [Background] Sheng L, Silvestrin T, Zhan J, Wu L, Zhao Q, Cao Z, Lou Z, Ma Q. Replacement of severely traumatized teeth with immediate implants and immediate loading: literature review and case reports. Dent Traumatol. 2015 Dec;31(6):493-503. doi: 10.1111/edt.12201. Epub 2015 Jul 14. PMID 26176171